CLINICAL TRIAL: NCT00062465
Title: A 24-Week, Double Blind, Randomized Study to Determine the Effects of 24 Weeks of Dosing With Tripterygium Wilfordii Hook F (TwHF) or Sulfasalazine, in Subjects With Active Rheumatoid Arthritis
Brief Title: Treating Rheumatoid Arthritis With Tripterygium Wilfordi Hook F or Sulfasalazine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030208; 03-AR-0208
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Rheumatoid Arthritis
Keywords: DMARD; Clinical Trial; Thunder God Vine; Chinese Herb; Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: TwHF

SUMMARY:
Various forms of the plant extract Tripterygium wilfordi Hook F (TwHF) have been used in China as a remedy for inflammatory diseases, including rheumatoid arthritis. The purpose of this study is to investigate how tolerable, safe, and effective TwHF is for patients with rheumatoid arthritis. Investigators will compare the therapeutic effects of TwHF with Sulfasalazine, an FDA-approved drug for arthritis.

Participants in this 24-week study must have had active rheumatoid arthritis for at least six months. Approximately 120 patients will participate. Participants will be assigned to one of two drug-treatment groups, TwHF or Sulfasalazine. They will be given the study drug at each of six clinic visits and will be asked to take two capsules three times each day with meals and water. During the clinic visits, investigators will obtain multiple blood samples; give physical exams; assess swollen, tender, and painful joints; and administer x-rays.

Study participants will be compensated up to $260 for their involvement in this study.

DETAILED DESCRIPTION:
This is a multi-center, randomized, active treatment controlled phase II study in patients with either new onset or therapy resistant rheumatoid arthritis (RA). This study will be conducted at 7 sites with NIAMS being the coordinating center and 6 external centers. Tripterygium wilfordii Hook F (TwHF) is a traditional medicinal plant that is and has been used in China for many years to treat inflammatory conditions including RA. This study we will be testing if a standardized plant extract from the roots of TwHF is superior to Sulfasalazine in improving the signs and symptoms in subjects with RA, as assessed by the ACR 20 criteria. Those subjects, who qualify for the study, will be allowed to continue on stable doses of NSAID therapy and/or low dose corticosteroids but will discontinue any DMARDs, or biologicals prior to the start of the study. Study subjects will then be randomized to receive either TwHF or Sulfasalazine and subjects will remain on double blind medication for 24 weeks. Patients will be assessed at baseline, 2 weeks and every 4 weeks thereafter using a standardized joint exam, questionnaires and laboratory measures for inflammation. ACR 20 responses will be calculated at each visit and compared in both groups at the end of evaluation at 24 weeks. Safety will be monitored throughout the trial. This is the first study that compares the extract of TwHF to a currently used DMARD in treating patients with RA and will help to define the role of new anti-inflammatory and possibly disease modifying agents in treating patients with RA.

ELIGIBILITY:
INCLUSION CRITERIA

Male and female outpatients between 18 and 75 years of age

Females must be of non-childbearing potential (post-menopausal, surgically sterilized or post hysterectomy) or using a double-barrier method of birth control for the duration of the study. A protocol acceptable method of double barrier method of birth control includes any combination of two or three of the following: condom, spermicidal and diaphragm.

Documented diagnosis of rheumatoid arthritis of at least six (6) months duration, as defined by the American Rheumatism Association 1987 Revised Criteria

American Rheumatism Association Functional Class I, II, or III

Meet the criteria for (active disease) at both screening and baseline visits by achieving all of the criteria below:

6 or more painful/tender joints

6 or more swollen joints

Visual Analog Scale (VAS) for pain of at least 3 (on scale of 1-10, where 1 is mild)

C-reactive protein (CRP) greater than or equal to 0.6 mg/dl or ESR greater than 25 mm/hr.

Prior/Current Therapy:

A. Subjects must be either DMARD or biological anti-RA agent naive or have failed a DMARD/biological RA agent, other than sulfasalazine, and have stopped this DMARD/biological one (1) month prior to randomization unless they have a flare in disease activity upon discontinuing DMARD/biological therapy as part of this protocol. DMARDs include but are not limited to methotrexate, leflunomide, minocycline, hydroxychloroquine, gold, cyclosporine, and biologics include anti-TNF and anti-IL-1 agents.

B. Subjects may be taking NSAIDs, provided the dose and frequency have been stable for 30 days prior to randomization. However if the patient meets the flare criteria they can be enrolled even if they have not fulfilled the criteria of being on a stable dose of NSAIDs and steroids for 30 days prior to randomization. At the time of flare neither steroids nor NSAIDs can be increased.

C. Subjects may be taking corticosteroid therapy equivalent to prednisone less than or equal to 7.5 mg/day. This dose must be stable for at least 1 month prior to randomization. Subjects may not change the dose of their corticosteroid or receive intra-articular or intra-muscular injections of corticosteroids, within 1 month of randomization or during the study. Note section 9.3 of the protocol, Concomitant Medication, has been amended to read: If it is medically necessary a one joint steroid injection is acceptable. This must be noted on the CRF and the joint excluded from the joint count.

D. Subjects may not be taking other complementary and/or alternative medications for RA for the last 1-month prior to randomization.

Subjects must provide written informed consent prior to any study-related screening tests.

EXCLUSION CRITERIA

Subjects with RA for less than six months duration, or onset before age 16 (JRA)

Clinically significant, uncontrolled concurrent neurological, hematological, renal, hepatic, endocrine, pulmonary, or cardiovascular disease

Subjects with evidence of an active clinically important cardiovascular disease as evidenced by an ECG at screening

Concomitant therapy or therapy within the last 30 days with another investigational drug

Subjects with screening laboratory values that deviate from the upper or lower limits of normal by greater that the percentages listed below:

* Liver function tests: Total bilirubin above the upper limit of normal (ULN). AST, ALT, 1.5 X greater than ULN
* Hematology: Total white blood count (WBC) less than 3500mm3. Hemoglobin and hematocrit less than 10 g/dl or 30%, unless stable for at least 3 months), and platelet count less than 100K or greater than 750 K.
* Renal function tests: BUN or creatinine greater than 1.2 X above the ULN
* Urinalysis: On dipstick - Proteinuria / hematuria / leukocytes greater than trace.

Subjects with serological evidence of chronic hepatitis B (positive HbsAG) or hepatitis C (positive C Ab), HIV

Subjects with evidence of active peptic ulcer disease or who have a reliable positive history of gastrointestinal bleeding within the past five (5) years. Any recurrent or history of an intestinal disorder that may interfere with the proper absorption of the drug

Pregnant women or nursing mothers

Subjects who plan to donate blood or blood products during the study or within 30 days following the last study visit.

One re-screening to meet criterion 6.1.5 will be allowed. Multiple screenings, beyond one for failure to meet criterion 6.1.5 are not allowed (at either screening or baseline).

Abuse of alcohol or drugs. The subject should not consume more than 2 units of alcohol per day. (A unit of alcohol is considered: 12 oz of beer, 6 oz of wine or 1 oz of spirits). This is on a per day basis and not the average for the week.

Subjects with a sulfonamide allergy

Subjects who have known G6PD deficiency

Subjects who are unable or unwilling to follow the protocol

Recent major trauma or major surgery or serious infection

Subjects who started but left, or were dropped out of this study, for any reason (subjects who left or are dropped will not be replaced).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157
Dates: Start 2003-06; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Tao X, Cai JJ, Lipsky PE. The identity of immunosuppressive components of the ethyl acetate extract and chloroform methanol extract (T2) of Tripterygium wilfordii Hook. F. J Pharmacol Exp Ther. 1995 Mar;272(3):1305-12. PMID 7891348
- [Background] Tao X, Cush JJ, Garret M, Lipsky PE. A phase I study of ethyl acetate extract of the chinese antirheumatic herb Tripterygium wilfordii hook F in rheumatoid arthritis. J Rheumatol. 2001 Oct;28(10):2160-7. PMID 11669150